CLINICAL TRIAL: NCT06855667
Title: Efficacy and Safety of Therapeutic Plasma Exchange vs Standard Medical Therapy in Severe Autoimmune Hepatitis: A Pilot Randomized Controlled Study
Brief Title: Efficacy and Safety of Therapeutic Plasma Exchange vs Standard Medical Therapy in Severe Autoimmune Hepatitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AIH-02
Record Dates: First submitted 2025-02-17; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Plasma Exchange; Steroids; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma Exchange (Experimental): 3 to 5 sessions +Steroids
  Interventions: Biological: Plasma Exchange; Drug: Steroid
- Standard Medical Treatment (Active Comparator): Steroids + Nutrition
  Interventions: Drug: Steroid; Dietary Supplement: Diet

INTERVENTIONS:
Biological: Plasma Exchange — 3 to 5 sessions alternate day
  Arms: Plasma Exchange
Drug: Steroid — Steroid
Dietary Supplement: Diet — Diet
  Arms: Standard Medical Treatment

SUMMARY:
Autoimmune hepatitis (AIH) is a chronic inflammatory liver disease that can lead to cirrhosis and liver failure. AIH can present in all ages, races, and ethnicities, but it mostly affects women. As a heterogeneous disease, AIH presents variably in different patients, making diagnosis and treatment a challenge.It is associated with varied clinical presentations and natural history and somewhat unpredictable treatment responses. Steroids and immunosupressants are main stay of treatment.In acute severe presentations corticosteroid response rates are more variable.According to treatment guidelines if patients fail to respond to corticosteroids, Liver transplant is the only option. But Liver transplant is not feasible in all situations such as limited donor availability.Plasma exchange is associated with a reduction in levels of pro-inflammatory cytokines,DAMPs, and bacterial endotoxins and increase in the levels of anti-inflammatory cytokines.Plasma exchange has reportedly been used for acute presentations of AIH but there are few trials which prove its independent benefit and role in influencing transplant free survival.The study aims at proving the efficacy of Plasma exchange as a bridge between steroid therapy and Liver transplant.It includes the patients with acute severe autoimmune hepatitis .One group of patients are taken up for plasma exchange sessions and compared with the other group started on high dose of steroids and they will be observed for 28 days and are assessed for transplant free survival and efficacy of plasma exchange in reducing transaminitis and Bilirubin levels.

DETAILED DESCRIPTION:
* Study population: Patients presenting with severe autoimmune hepatitis and MELD>24 with no liver transplant option.
* Study design: A Pilot Randomised control trial
* Study period: 2 year
* Sample size:
* There is no studies of PE in severe AIH, assuming effect of PE in ACLF group
* Survival rate with plasma exchange was assumed to be 60 % and 20 % without PE.
* Further assuming 95% power and alpha 5 %.
* We need to enroll 46 cases i.e. 23 in each group
* Further assuming % defaulter rate, it is further decided to enroll 25 cases in each group.
* Patients will be randomly allocated in 2 groups by 1:1 block randomisation and will be implemented by IWRS facility taking block size 10.
* Monitoring and assessment: All patients would undergo vital and baseline parameter screening before randomization. Based on randomization they will receive either steroid or plasma exchange followed by steroid.
* Interim analysis would be done to check efficacy and safety of TPE in severe autoimmune hepatitis.
* Adverse effects:

Therapeutic Plasma Exchange is associated with risk of adverse events like infections,Fluid overload or circulatory insufficiency, Hypersensitivity to blood products.

- Stopping rule: Study will be stopped in case of life- threatening events occur in patient after randomisation

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Acute severe autoimmune hepatitis with MELD >24
3. No liver transplant option < 28 days.
4. -ACLF + Non ACLF
5. Auto immune hepatitis: Diagnosis by simplified AIH score ≥6

Exclusion Criteria:

1. Patients with Active sepsis
2. Patients with Active bleeding
3. Patients allergic to FFP and blood products
4. Patients with unstable hemodynamics ( eg:BP<90/60 mmhg,HR >100bpm)
5. Patients with post renal obstructive AKI, AKI suspected due to glomerulonephritis, interstitial nephritis or vasculitis based on clinical history and urine analysis
6. Pregnancy related liver failure
7. Comorbidities associated with poor outcome (Extrahepatic neoplasia, severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease)
8. Refusal to participate in the study
9. Patients who are eligible to transplant
10. Patients who received steroids or on steroids last 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with change in AST,ALT,Bilirubin | 28 days

SECONDARY OUTCOMES:
Liver transplant free survival at 28 days. | 28 days
Development of adverse event due to TPE | 28 days
Number of patients with development of clinical infection during study period | 28 days
  Clinical infections includes pneumonia, SBP,UTI,soft tissue infections,blood stream infections.
Mortality during hospital stay | 28 days
Change in grade of HE, grade of ascites (both ascites and HE if present). | 28 days
Frequency of decompensation events on follow up period. | 28 days
Infections at 28 days | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided